CLINICAL TRIAL: NCT04755933
Title: A Randomised Controlled Trial of an Online Intervention to Prevent Anxiety in the Children of Anxious Parents
Brief Title: Parenting With Anxiety: Helping Anxious Parents Raise Confident Children
Acronym: PWA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sussex (Other)
Collaborators: Kavli Trust (Unknown); Brighton & Sussex Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ER/SC430/1
Record Dates: First submitted 2021-02-02; First posted 2021-02-16 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Child Anxiety; Parent Anxiety; Parental Wellbeing; Child Wellbeing
Keywords: Parenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): An online learning tool, designed to helps parents develop a calm, consistent behaviour management style, whilst learning skills to discourage children's avoidance.
  Interventions: Behavioral: Raising Confident Children Course
- Control (No Intervention): The participants in the control arm will not receive access to the online course, but will complete the same sets of questionnaires at each of the timepoints.

INTERVENTIONS:
Behavioral: Raising Confident Children Course — An online learning tool consisting of 8 different modular components, designed to reduce the transmission of anxiety from parents to children. The modular components include: a core starter about anxiety, the role of avoidance, using play to develop childrens confidence, using Emotion Coaching with children, managing difficult behaviour, the role of sleep, exercise and diet, reducing overprotection, modelling confident behaviour and managing difficult behaviour.
  Arms: Intervention

SUMMARY:
This is a randomised controlled trial of an intervention to reduce symptoms of anxiety in the children of anxious parents. Parents will participate in an online intervention which helps them develop a calm, consistent, behaviour management style. The parents will be randomised to the intervention or a control group with no intervention. The intervention itself will undergo a component analysis to determine whether some modules are more effective than others.

DETAILED DESCRIPTION:
The study is an online course (derived from an existing evidence-based face-to-face workshop designed and evaluated by the C.I) which aims to reduce symptoms of anxiety in the children of anxious parents. It is a learning tool to help parents to understand the basic processes involved in children's anxiety, to develop a calm, consistent, behaviour management style and to learn skills for responding to difficult emotion in their children.

The whole study takes place online, allowing the participants to sign up, run through some brief eligibility questions, read the study information and provide consent.

Once enrolled in the study, there is a series of baseline questionnaires. The participant also has the option to nominate someone who also knows their child well (e.g. a co-parent, a family member or close friend) to participate in the study with them and to complete a small number of questionnaires. This will help to give us a broader, more objective picture of the child, but is an optional part of the study. 48 hours later (to allow time for the participants to contact the co-respondent if they choose) the index participant will be randomised to one of two groups: either the intervention (the online course), or the control group where they do not receive the intervention.

Those in the intervention will be randomised to receive 8 out of 9 modules of the course, with a suggested time frame of one or two modules a week, each module taking about 30 minutes, with some home-practice tasks in-between.

Both the intervention group and the control group participants will be contacted again after 6 months to complete a set of follow-up questionnaires (similar to those completed at baseline). Depending on when each participant joins the trial, they may be contacted a third time towards the end of the life of the study, to complete another set of questionnaires,9-21 months after their first.

ELIGIBILITY:
Inclusion Criteria:

* Be a parent (any gender, adoptive/biological/step/foster/grandparent) aged 16+, of a child aged 2 to 11 years (inclusive). The index parent must have at least 50 days' contact with the index child per year and confirm that they see enough of the child to report on the child's current anxiety level.
* Index parent must be a UK resident.
* Self-report subjectively substantial levels of current or lifetime anxiety.
* Able to commit to completion of measures at (up to) three time points even if allocated to the control arm.

Exclusion Criteria:

* N/A

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3508 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in child anxiety | Baseline, 6 months, and up to 21 months.
  Measured using the Spence Children's Anxiety Scale (SCAS-P and Preschool SCAS if the child is aged 6 or under).
  SCAS-P: Minimum 0 Maximum 114. A higher total score is indicative of higher level of child anxiety. T scores used to indicate clinical levels of anxiety however this is a screen not a diagnostic instrument.
  SCAS Preschool: Minimum 0 Maximum 112. A higher total indicates a higher level of pre-school child anxiety. A score of 1SD above the mean for a subscale or the total score indicates clinical investigated would be warranted.

SECONDARY OUTCOMES:
Change in parent anxiety and parental wellbeing | Baseline, 6 months, and up to 21 months.
  Measured using Screen for Child Anxiety Related Emotional Disorder (SCARED-A): Minimum 0, Maximum 142. . Higher total score (>30) predictive of a current anxiety disorder. Higher subscale scores associated with elevated anxiety symptoms of clinically defines anxiety disorders.
Change in parent anxiety and parental wellbeing | Baseline, 6 months, and up to 21 months.
  Measured using Short Warwick Edinburgh Mental Wellbeing Scale. Minimum score 7. Maximum score 35. Raw scores converted into metric scores. Higher scores indicate higher positive mental wellbeing.
Change in child wellbeing and health | Baseline, 6 months, and up to 21 months.
  Measured using Pediatric Symptom Checklist (PSC-17). Minimum 0. Max 35. A higher score indicates a worse psychosocial functioning. Scores predictive of psychopathology at following levels: Internalizing score positive if ≥ 5 PSC-17 Externalizing score positive if ≥ 7 PSC-17 Attention score positive if ≥7 PSC-17 Total score positive if ≥15.
Change in child wellbeing and health | Baseline, 6 months, and up to 21 months.
  Measured using EQ-5D-Y Proxy. Minimum 11111 Maximum 33333. A higher score indicates a worse health status.
Change in anxiogenic parenting behaviours | Baseline, 6 months, and up to 21 months
  Measure using Comprehensive Parenting Behaviour Questionnaire (CPBQ). Minimum 104. Maximum 520. The scale is split into broad dimensions, subscales and sub subscales. Higher scores are associated with greater level of parenting behaviour under investigation in the given subscale: both positive (e.g. warmth) and challenging (e.g. overprotection).
Change in anxiogenic parenting behaviours | Baseline, 6 months, and up to 21 months
  Measured using a parenting experience scale (constructed specifically for this study, divided into 8 modules).
  Core: Min 1 Max 5. Higher score = Positive. Module A: Min 1 Max 5. Higher score = Positive (Q2: R scored). Module B: Min 1 Max 5. Higher score = Positive (all are R scored). Module C: Min 1 Max 5. Higher score = Positive. Module D: Q1, Q3, Q4: Min 1 Max 5. Higher score = Positive (Q4: R scored). Module D Q2: Min 1 Max 5. Higher score = Positive. Module E: Min 1 Max 4. Higher score = Negative (Q3: R scored). Module F: Min 1 Max 5. Higher score = Positive (Q1 and Q4: R scored). Module G Q1: Min 1 Max 5. Higher score = Positive (Q1: R scored). Module GQ2: Min 3 Max 5: Higher score Negative (Note: Both ends of the scale are maladaptive). Module G Q3: Min 1 Max 5. Higher score = Negative.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Cartright-Hatton, Principal Investigator — University of Sussex
Locations (1):
- University of Sussex, Brighton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will not be shared on an individual basis. Anonymised study data will be archived at the end of the study through the University of Sussex data repository, Figshare.

REFERENCES:
- [Derived] Dunn A, Alvarez J, Arbon A, Bremner S, Elsby-Pearson C, Emsley R, Jones C, Lawrence P, Lester KJ, Morson N, Simner J, Thomson A, Cartwright-Hatton S. Effectiveness of an unguided modular online intervention for highly anxious parents in preventing anxiety in their children: a parallel group randomised controlled trial. Lancet Reg Health Eur. 2024 Sep 4;45:101038. doi: 10.1016/j.lanepe.2024.101038. eCollection 2024 Oct. PMID 39291249
- [Derived] Dunn A, Alvarez J, Arbon A, Bremner S, Elsby-Pearson C, Emsley R, Jones C, Lawrence P, Lester KJ, Majdandzic M, Morson N, Perry N, Simner J, Thomson A, Cartwright-Hatton S. Effectiveness of a Web-Based Intervention to Prevent Anxiety in the Children of Parents With Anxiety: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Nov 10;11(11):e40707. doi: 10.2196/40707. PMID 36355406